CLINICAL TRIAL: NCT06932900
Title: French Translation and Validation of the Banff Patellar Instability Instrument 2.0
Brief Title: French Version of the Banff Patellar Instability Instrument 2.0
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, François Vézina, orthopaedic surgeon, Université de Sherbrooke
Other Study IDs: 2022-4329
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Patellar Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- validation: person with patellar instability that will respond to the questionnaires

SUMMARY:
There are several treatment options for patellofemoral instability, but no established guidelines currently exist. An important step toward developing a consensus is to examine the influence of each intervention through the collection of both subjective and objective outcomes.

Most outcome measures commonly used for knee pathologies are primarily designed to monitor degenerative conditions (e.g., osteoarthritis) or ligamentous instability (e.g., anterior cruciate ligament rupture). Very few questionnaires are specific to patellar instability, a condition characterized by distinct signs and symptoms compared to other knee disorders.

The Banff Patellar Instability Instrument (BPII) was developed with this gap in mind, in accordance with the Consensus-based Standards for the Selection of Health Measurement Instruments (COSMIN) criteria. This condition-specific tool is designed to subjectively assess the functional impact of patellofemoral instability on patients' quality of life, which is the most important factor in evaluating treatment success.

Currently, there is no validated French-language outcome measure specific to patellofemoral instability. To improve patient care, the availability of such a validated tool in French is essential, both for clinical use and for conducting future research.

To address this issue, the primary objective of this study is to translate the Banff Patellar Instability Instrument 2.0 (BPII 2.0) into French, following the three-step process described in the IQOLA project and in accordance with the guidelines outlined by the American Academy of Orthopaedic Surgeons (AAOS), and to evaluate its validity in a French-speaking population.

Research Question Is the French version of the BPII 2.0 a valid tool to assess function in French-speaking patients diagnosed with patellofemoral instability?

Specific Objectives

To translate the Banff Patellar Instability Instrument 2.0 into French using a dual forward-backward translation process.

To evaluate the psychometric properties of the French version of the BPII 2.0, including its reliability and validity.

DETAILED DESCRIPTION:
To address our primary outcome described above, an analytical observational design has been chosen as no intervention is applied to the subjects under study. The prospective study will confirm our hypothesis for objective 2, which is the validation of the questionnaire translated into French.

Study Population and Sample

The target population for this study consists of all patients with patellofemoral instability whose native language is French. Due to the difficulty of accessing such a large pool of patients, we will use an accessible population, specifically all French-speaking patients with patellofemoral instability who consult with an orthopedic surgeon at the Centre Hospitalier Universitaire de la Santé (CHUS) in Fleurimont, Hôtel-Dieu Hospital, or the Shriners Hospitals for Children - Canada in Montreal.

Selection Criteria

For the pre-test during the translation stage, all individuals aged 14 years or older, whose native language is French, are being followed for a knee condition at the CHUS outpatient clinic or Hôtel-Dieu Hospital, and who are willing to participate in the validation of the BPII 2.0 questionnaire translation will be included. No specific diagnosis of patellofemoral instability is required.

For the validation stage, the project will be presented to all patients at the CHUS Fleurimont, Hôtel-Dieu Hospital, or Shriners Hospitals for Children in Montreal, who are diagnosed with patellofemoral instability by an orthopedic surgeon and meet the criteria listed below. Patients with other pathologies of the affected lower limb or disease progression will be excluded to avoid confounding factors impacting functional quality of life. Also, those answering fewer than 19 questions will be excluded, as this corresponds to an invalid score according to studies of the test in English (4,6). To improve recruitment rates, we are making the project multicentric, and the orthopedic department at Shriners Hospitals for Children in Montreal will participate in the validation phase.

Inclusion Criteria

Patients aged 14 years and older with a new diagnosis of patellofemoral instability confirmed by an orthopedic surgeon

With conservative and/or surgical treatment

Patients fluent in both oral and written French

Exclusion Criteria

Patients who are unable to understand and/or respond to the questionnaire

Patients with another diagnosis or knee pathology under study (e.g., complex ligament tear, gonarthrosis)

Patients with another diagnosis or lower limb pathology under study with secondary functional impairment (e.g., coxarthrosis)

Patients with a change in the condition of the affected lower limb

Exclusion from test-retest reliability calculations if symptoms of patellofemoral instability worsen or new involvement of this lower limb occurs between T0 and T1

Exclusion from the response to change calculation if new involvement of the lower limb (e.g., ipsilateral lower limb trauma) occurs after treatment, i.e., between T0 and T2

Patients answering fewer than 19 questions (out of 23)

Sampling

To recruit eligible patients for the study, we will proceed with a non-probability convenience sampling approach.

For the first stage of translation (pre-test), all individuals who meet the criteria listed above will be included. For the second stage of validation, we will present the study to all patients who meet the selection criteria and present at the outpatient clinics of CHUS, Hôtel-Dieu Hospital, and Shriners Hospitals for Children in Montreal. This approach does not guarantee the representativeness of the population with patellofemoral instability, but it will not impact the validation of the functional measurement tool. This method will allow us to recruit a sufficient number of patients within a reasonable time frame. There are no confounding factors involved in the sampling of the population, as the goal of this study is the qualitative validation of the test, not measuring the treatment effect.

Recruitment

Participant recruitment will be on a voluntary basis. For the pre-test translation stage, patients will be recruited at the orthopedic outpatient clinic of CHUS Fleurimont or Hôtel-Dieu Hospital. For the validation stage, at the time of diagnosis, the orthopedic surgeon or resident at CHUS Fleurimont or Hôtel-Dieu Hospital who confirms patellofemoral instability will introduce the research project to the patient and verify if they meet the established selection criteria. If available at the participating center, the orthopedic surgeon or resident will have the patient sign a contact authorization form, if the research assistant is unavailable, to indicate whether the patient agrees to meet with the research assistant (Appendix 3). If the patient agrees to meet the research assistant, they will receive all relevant information about the research project. Together with the research assistant, the patient will be able to freely consent to their inclusion or exclusion from the research project by signing the informed consent form (refer to the consent form for the research project). In the case that the contact authorization form is unavailable, the research assistant will approach the patient after confirmation of the patellofemoral instability diagnosis during their clinic appointment.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with patellar instability with conservative or surgical treatment
* fluent in both spoken and written French

Exclusion Criteria:

* Patients who are unable to understand and/or respond to the questionnaire
* Patients with another diagnosis or knee pathology under study (e.g., complex ligament tear of the knee, gonarthrosis)
* Patients with another diagnosis or lower limb pathology under study with secondary functional impairment (e.g., coxarthrosis)
* Patients with a change in the condition of the lower limb under study a. Exclusion from test-retest reliability calculations if symptoms of patellofemoral instability worsen or if there is new involvement of this lower limb between T0 and T1 b. Exclusion from response to change calculations if new involvement of the lower limb (e.g., ipsilateral lower limb trauma) occurs after treatment, i.e., between T0 and T2
* Patients answering fewer than 19 questions (out of 23 questions)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting at the CHUS in Sherbrooke or at the Schriners Hospital in Montreal for patellar instability
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Banff Patellar Instability 2.0 Index in French | Baseline, 1 week and 6 month post intervention
  Questionnaire. (0-100 (0 = Worst, 100 = Best))
Questionnaire Anterior Knee Pain Scale (Kujala) | Baseline and 6 month post intervention
  Questionnaire. (0-100 (0 = Worst, 100 = Best))
Socio-Demographic | Baseline
  Age, Sex, Time since symptoms, Scolarship, Nationality

CONTACTS AND LOCATIONS:
Overall Officials: François Vézina, Doctor, Principal Investigator — Université de Sherbrooke
Locations (1):
- CIUSSS de l'Estrie-CHUS, 3001, 12e Ave Nord, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
This was not mention in the consent form as required in our REB. We could share the data on demand but not on public registry